CLINICAL TRIAL: NCT03427489
Title: A Biorepository for Discovering Novel Biochemical and Genetic Markers of Coronary Heart Disease in Qatar (QCBio)
Brief Title: A Biorepository for Coronary Heart Disease in Qatar
Acronym: QCBio
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dr. Ayman El-Menyar, Associate Professor, Hamad Medical Corporation
Other Study IDs: NPRP No. : 5 - 1024 - 3 - 225
Record Dates: First submitted 2018-01-01; First posted 2018-02-09 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: Biomarkers; Genetic Markers; Controls
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We intend to establish a DNA and plasma repository of 1000 Qatari CHD cases and 1000 ethnicity-matched controls (QCBio) to enable investigation of genomic and proteomic biomarkers for early detection and prognostication and to identify new targets for drug development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary heart disease: Qatari individuals presenting with or have a history of an acute coronary syndrome (myocardial infarction or unstable angina) are being recruited as study subjects.
- Controls: Ethnicity-matched individuals without history of CHD such as myocardial infarction or prior PCI are being recruited as controls.

SUMMARY:
Coronary heart disease (CHD) poses a major health burden in the Gulf countries. It is the leading cause of mortality and morbidity in the world and poses an enormous societal burden in the Gulf countries. Early detection of disease is imperative to reduce the health care burden and financial costs associated with CHD. Knowledge of novel genetic and proteomic markers of CHD will provide more precise estimates of risk while defining the pathways important in individual patients, revealing new targets for intervention, and ultimately enabling an individualized approach to care.

To translate recent advances in genomics and proteomics into clinical practice, these newly discovered biomarkers will need to be evaluated in patients of diverse ethnic groups with varying characteristics, environmental factors, and medication use. The investigators propose to establish a biorepository of plasma and Deoxyribonucleic acid (DNA) linked to demographic and clinical variables to facilitate biomarker studies of CHD risk, progression, and outcome. The overarching goal in developing the Qatar Cardiovascular Biorepository (QCBio) is to create a resource that fosters research aimed at identifying novel biochemical and genetic markers of CHD. A biorepository with linkage to clinical data will also provide an invaluable resource for cardiovascular research, including genomic and proteomic studies of CHD and development of biomarkers for early detection of disease and personalized drug therapy (pharmacogenetics and pharmacoproteomics).

DETAILED DESCRIPTION:
INTRODUCTION:

Prediction of Coronary heart disease (CHD) events is based on conventional risk factors for atherosclerosis such as age, sex, blood pressure, diabetes, lipid levels, and smoking status. Because these risk factors are prevalent in much of the population, available risk prediction algorithms lack desired sensitivity and specificity. For instance, Cooper et al showed that the algorithms correctly predicted just ~11% of the CHD events occurring within 10 years. Thus, there is an urgent need to develop and validate new biomarkers for early detection of disease and more accurate risk stratification. According to the World Health Organization (WHO) estimates, cardiovascular disease will be the leading cause of morbidity and mortality by the year 2020. Developing countries including the Gulf States will be the major contributors to this increased death and disability. A recent report by McKinsey & Company forecast that the Gulf region will face an unparalleled and unprecedented rise in demand for health care over the course of the next two decades, with an estimated total health care spending of US$ 60 billion in 2025, up from US$ 12 billion today.

Knowledge of novel genetic and proteomic markers will provide more precise estimates of risk while defining the pathways important in individual patients, revealing new targets for intervention, and ultimately enabling an individualized approach to care. A biorepository of Deoxyribonucleic acid (DNA), serum, and plasma samples will enable investigation of the pathogenesis of CHD in Qatari adults, and provide an invaluable resource for preventive cardiovascular research and development of biomarkers for early detection of CHD.

SIGNIFICANCE Significant recent progress has been made in identifying genetic susceptibility variants as well as circulating proteomic markers of atherosclerotic vascular disease. However, the generalizability of these results to patients belonging to diverse ethnic groups is unclear. To translate recent advances in genomics and proteomics into clinical practice, these newly discovered biomarkers will need to be evaluated in patients of diverse ethnic groups with varying characteristics, environmental factors, and medication use. The investigators propose to establish a biorepository of plasma and DNA linked to demographic and clinical variables to facilitate biomarker studies of CHD risk, progression, and outcome. The overarching goal in developing the Qatar Cardiovascular Biorepository (QCBio) is to create a resource that fosters research aimed at identifying novel biochemical and genetic markers of CHD.

RESEARCH DESIGN AND METHODS:

The investigators are leveraging the following resources available for this proposal:

1. The infrastructure and patient referral patterns of the cardiac catheterization laboratory at Hamad Hospital, Doha, Qatar, where several thousand patients are seen annually for coronary angiography and percutaneous coronary intervention;
2. The Electronic Medical Record (EMR) at Hamad Hospital that includes risk factors, drug therapy, relevant laboratory data, and vital status; and
3. A multidisciplinary investigative team with significant experience and expertise in biorepository science, including ethical, legal, and social implications (ELSI), laboratory information management systems, informatics, and mining of the EMR to annotate biospecimen with relevant clinical covariates.

SPECIFIC AIMS AND OBJECTIVES:

1. Establish a DNA and plasma biorepository (QCBio) of Qatari CHD cases and ethnicity-matched controls to enable investigation of genomic and proteomic biomarkers for early detection and prognostication as well as identification of new targets for drug development.
2. Annotate the biorepository with a) demographic, laboratory, and clinical variables derived from the EMR using electronic phenotyping algorithms, and b) detailed information regarding history of cardiovascular diseases and risk factors derived from surveys of the study subjects.
3. Develop processes to promote use of the biorepository by Qatari investigators by facilitating access to the biorepository for biomarker research, while maintaining the highest ethical standards with emphasis on patient confidentiality and stewardship of the biospecimens.
4. Tracking Recruitment: A Patient Numbering Program (PNP) is being used to de-identify subjects enrolled in the study and track patient recruitment. The program contains demographic information and an assigned Personal Identification Number (PIN) for each participant.

Consenting: Potential subjects are being identified by the study coordinators after review of catheterization laboratory (Cath lab) and blood bank schedules. The study coordinator is explaining the consent form and the study questionnaire to each participant. Wherever possible, the investigators are attempting to collect blood specimens in the fasting state before the receipt of any treatment and avoid the burden of additional venipuncture. For those eligible ones, the study coordinator will provide the details regarding the objectives of the study, risks and potential benefits from participation, the storage, future use and privacy of the samples. In addition, the study coordinator is informing the participants about the lack of immediate benefit for health and their right to withdrawal from the study any time after consenting.

Collection and Processing of Blood Samples: Twenty-five milliliter of blood is being obtained at the time of a procedure in the Cath lab, during admission in the Coronary care unit (CCU) or at the time of the blood donation. Samples are collected from the special study area close to the Cath Lab/CCU and the Blood Bank, respectively. Blood is being drawn into the appropriate collection tubes, labeled with a hospital generated barcode Identification number, and sent to the Molecular Genetics laboratory.

Freezer Monitoring: All freezer temperatures are being monitored round the clock by a combination of project management facilities and Hamad Medical Corporation (HMC) Security.

Quality Assurance: Accurate sample handling is being achieved by adherence to Standard Operating Procedures (SOPs) by following general laboratory quality assurance and control standards.

Specimen Tracking: Sample tracking will be accomplished by a Laboratory Information Management System (LIMS) program that is currently being used by the Lead PI's research group.

Patient Confidentiality: The investigators will use informatics and data security features to maintain patient confidentiality. The Patient Numbering Program (PNP) will be used to de-identify patients enrolled in QCBio and to track patients after recruitment.

Ethical, Legal, and Regulatory Issues in DNA Biorepositories: The consent form is including separate check-off boxes to seek permission for the collection of plasma and DNA use in studies of diverse diseases, and the transmittal of specimens to collaborating investigators. Banking of biospecimens raises new concerns regarding a patient's privacy and consent.

Informatics: Informatics and data security are critical components to a biorepository and key to leveraging the power of biorepositories. QCBio will be linked to several databases.

Study Questionnaire: The investigators are using a questionnaire to collect information regarding sociodemographic information, cardiovascular history, physical activity, lifestyle, past medical information and family history. Data will be extracted from the questionnaire by scanning or manual entry.

Annotation of Specimens with Clinical Data: The investigators are using the Hamad hospital EMR viewer in addition to the laboratory databases to annotate the biorepository with relevant clinical variables.

Ascertaining Risk Factors: The investigators are ascertaining conventional cardiovascular risk factors, including hypertension, diabetes, and dyslipidemia. The EMR and survey data will be used to establish presence of the following risk factors for atherosclerosis: smoking, diabetes, hypertension, dyslipidemia, and obesity. The investigators are using targeted manual review of paper records and EMR in tandem with access to electronic data sets for laboratory values, medications, and diagnosis codes.

Biospecimen Management and Access to Biorepository: The investigators will develop protocols to enable investigators to leverage the datasets associated with specimens, ensure compliance with regulatory guidelines, encourage collaboration between Qatar, Gulf, and Mayo investigators, and improve research productivity. The investigators will provide a flexible, robust, secure, and validated information management workspace program to manage biospecimens. Banked specimens will be available for researchers whose protocols have been approved by the IRB and prioritized by the Scientific Review Panel.

Tracking Specimen Use: To maximize the use of the biospecimens, the investigator will use LIMS to track all the specimens received by allotting unique identification for all input (sample tubes) and output (DNA/plasma/white cell) tubes and record the sample movement, processing, creation, and consumption. A designated computer analyst will maintain and manage the system.

Access to Information: Only members of the research team will have access to the research data. Participants will be identified by code numbers only in the database and in transcripts; all data are tracked in databases by anonymous but linkable study numbers. No identifiable information will be released outside the study.

Strategy for Project Continuation: The long-term goal of the investigative team is to create a resource that enables discovery of genetic susceptibility variants and novel circulating markers of CHD, thereby allowing individualized assessment of risk for CHD, a leading cause of death and morbidity in Qatar. Creation of the biorepository is the first necessary step to understand genomic and proteomic of CHD in Qatari individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects: History or clinical diagnosis of Acute Coronary Syndrome
* Controls: No history of Coronary Heart disease.

Exclusion Criteria:

* Chronic or infectious disease
* Vulnerable populations (Children, prisoners, cognitive impairment)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Qatari individuals who present with or have a history of an acute coronary syndrome (myocardial infarction or unstable angina) are being recruited as study subjects from the coronary catheterization laboratory (Cath Lab) and the coronary care unit.
  Ethnicity-matched controls are being recruited from the blood bank where individuals typically undergo screening by means of questionnaires and those with chronic or infectious disease are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Identification of genetic variants associated with CHD in Qatari Individuals using whole genome sequencing on the 2000 samples stored at the genetic biorepository over 3 years. | Three years
  QCBio will create an unparalleled and unique resource for conducting genomic and studies to identify and validate biomarkers for diagnosis, prognostication, and response to therapy, in Qataris patients who have CHD or at risk

SECONDARY OUTCOMES:
Identification of circulating markers using plasma proteomic and metabolomic analysis in 2000 Qatari individuals with and without CHD. | Three years
  Candidate approach with markers in etiologic pathways of atherosclerosis including inflammation, lipids, hemodynamic regulation, thrombosis and metabolism in addition to Agnostic approach using plasma metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Iftikhar Kullo, Principal Investigator — Mayo Clinic College of Medicine; Ayman El-Menyar, Principal Investigator — Hamad Medical Corporation; Jassim Al Suwaidi, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Khoja T, Rawaf S, Qidwai W, Rawaf D, Nanji K, Hamad A. Health Care in Gulf Cooperation Council Countries: A Review of Challenges and Opportunities. Cureus. 2017 Aug 21;9(8):e1586. doi: 10.7759/cureus.1586. PMID 29062618
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Kullo IJ, Ballantyne CM. Conditional risk factors for atherosclerosis. Mayo Clin Proc. 2005 Feb;80(2):219-30. doi: 10.4065/80.2.219. PMID 15704777
- [Background] Cooper RS, Psaty BM. Should ethnicity serve as the basis for clinical trial design? Diversity and inclusiveness should remain the guiding principles for clinical trials. Circulation. 2005 Dec 6;112(23):3660-5; discussion 3665-6. No abstract available. PMID 16333866
- [Background] Kullo IJ, Cooper LT. Early identification of cardiovascular risk using genomics and proteomics. Nat Rev Cardiol. 2010 Jun;7(6):309-17. doi: 10.1038/nrcardio.2010.53. Epub 2010 May 4. PMID 20440292
- [Background] Morrison AC, Bare LA, Chambless LE, Ellis SG, Malloy M, Kane JP, Pankow JS, Devlin JJ, Willerson JT, Boerwinkle E. Prediction of coronary heart disease risk using a genetic risk score: the Atherosclerosis Risk in Communities Study. Am J Epidemiol. 2007 Jul 1;166(1):28-35. doi: 10.1093/aje/kwm060. Epub 2007 Apr 18. PMID 17443022
- [Background] Khoury MJ, Jones K, Grosse SD. Quantifying the health benefits of genetic tests: the importance of a population perspective. Genet Med. 2006 Mar;8(3):191-5. doi: 10.1097/01.gim.0000206278.37405.25. No abstract available. PMID 16540755
- [Background] Cortese DA. A vision of individualized medicine in the context of global health. Clin Pharmacol Ther. 2007 Nov;82(5):491-3. doi: 10.1038/sj.clpt.6100390. PMID 17952101
- [Background] Ginsburg GS, Burke TW, Febbo P. Centralized biorepositories for genetic and genomic research. JAMA. 2008 Mar 19;299(11):1359-61. doi: 10.1001/jama.299.11.1359. No abstract available. PMID 18349099
- [Background] Ding K, Kullo IJ. Genome-wide association studies for atherosclerotic vascular disease and its risk factors. Circ Cardiovasc Genet. 2009 Feb;2(1):63-72. doi: 10.1161/CIRCGENETICS.108.816751. No abstract available. PMID 19750184
- [Background] Kim CX, Bailey KR, Klee GG, Ellington AA, Liu G, Mosley TH Jr, Rehman H, Kullo IJ. Sex and ethnic differences in 47 candidate proteomic markers of cardiovascular disease: the Mayo Clinic proteomic markers of arteriosclerosis study. PLoS One. 2010 Feb 5;5(2):e9065. doi: 10.1371/journal.pone.0009065. PMID 20140090
- [Background] Evans BJ, Meslin EM. Encouraging translational research through harmonization of FDA and common rule informed consent requirements for research with banked specimens. J Leg Med. 2006 Jun;27(2):119-66. doi: 10.1080/01947640600716366. No abstract available. PMID 16728351
- [Background] Kullo IJ, Fan J, Pathak J, Savova GK, Ali Z, Chute CG. Leveraging informatics for genetic studies: use of the electronic medical record to enable a genome-wide association study of peripheral arterial disease. J Am Med Inform Assoc. 2010 Sep-Oct;17(5):568-74. doi: 10.1136/jamia.2010.004366. PMID 20819866